CLINICAL TRIAL: NCT01161056
Title: Genes and Phenotype (GAP) A National Resource for Genotype-Phenotype Studies of Immunological and Inflammatory Pathways
Acronym: GAP
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Peter Gregersen, Center Head, Northwell Health
Other Study IDs: 09-081A; 1RC2AR059092-01 (NIH)
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Immune System Diseases
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Blood sample will be processed to isolate DNA and peripheral blood mononuclear cells, which will be stored in our Biorepository.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Control Group

SUMMARY:
The purpose of this study is to enrol generally healthy adults, who are asked to provide a blood sample, to study how the immune system works.

DETAILED DESCRIPTION:
The primary purpose of this research is to develop a better understanding of how the immune system works. By studying immune function in many people, we will be able to determine the range of normal variation.

The second purpose is to enroll people who are willing to serve as comparisons in future research studies into the Genotype and Phenotype Research Registry (GAP Registry).

Volunteers are asked to provide information on age, ethnicity and medical history. Volunteers are asked to provide a blood sample of up to 100cc and allow us to contact you about additional studies.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* Generally healthy

Exclusion Criteria:

* History of autoimmune disease
* History of chronic immunodeficiency or chronic viral infections such as Epstein Barr virus, hepatitis or HIV
* Currently undergoing treatment for cancer
* Current treatment with immuno-suppressant drugs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2009-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of healthy participants enrolled | 5 years
  This is a registry to enroll healthy individuals who are interested in being contacted about research studies they can participate in as a healthy control

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gregersen, MD, Principal Investigator — Northwell Health
Locations (1):
- The Feinstein Institute for Medical Research, Manhasset, New York, United States